CLINICAL TRIAL: NCT01272843
Title: Physiological Magnetic Resonance Imaging (MRI) to Improve Carotid Endarterectomy Outcomes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Bradley J MacIntosh, Scientist, Sunnybrook Health Sciences Centre
Other Study IDs: CEACOG2011
Record Dates: First submitted 2011-01-06; First posted 2011-01-10 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2010-12

CONDITIONS: Carotid Stenosis; Hypoperfusion; Transient Ischemic Attack
MeSH Terms: conditions — Carotid Stenosis; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Carotid endarterectomy patients
- Lumbar stenosis laminectomy patients

SUMMARY:
The carotid arteries are blood vessels in the neck that supply blood to the brain. Carotid stenosis disease is defined as a narrowing of these arteries due to the build up of plaque. The plaque material can also break off and move into the brain. The resulting blockage of blood supply to a portion of the brain is what causes 80% of all strokes. One treatment option is to have surgery on the carotid artery and remove the plaque. This procedure is called a carotid endarterectomy (CEA). There is evidence that proves CEA reduces the risk of stroke. The objective of this research project is to determine who is most likely to benefit from CEA surgery.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 30 years of age
* Greater than grade 9 education level
* Mini-mental state exam (MMSE) greater than 19 for carotid stenosis patients

Exclusion Criteria:

* History of acute stroke
* History of current psychiatric disorder, such as depression or movement disorder
* Diagnosed Alzheimer's Disease or dementia

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Atherosclerosis is a major risk factor for ischemic cerebrovascular events such as stroke (Bots, Hoes et al. 1997). Carotid endarterectomy (CEA) and carotid stenting (CAS) are common surgical procedures aimed at reducing stroke risk. For individuals with symptomatic stenosis > 70%, CEA has a higher event-free survival compared to medical therapy (Barnett, Taylor et al. 1998) and is considered highly beneficial treatment (Rothwell, Eliasziw et al. 2003). To date, however, few studies have attempted to relate effects of the surgery to changes in brain physiology and function.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-03 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Functional MRI (fMRI) results will be used to calculate the activation-related hemodynamic response function (HRF) in patients undergoing carotid endarterectomy, which will be significantly reduced post-operative at 3 months follow-up. | Pre-operative, 3 months post-operative

SECONDARY OUTCOMES:
Dynamic intracranial angiography will be correlated with arterial arrival time (AAT) hemodynamic metric calculated from arterial spin labeling (ASL) perfusion MRI. | Pre-operatively, 3 months post-operatively

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Research Institute, Toronto, Ontario, Canada

REFERENCES:
- [Result] MacIntosh BJ, Filippini N, Chappell MA, Woolrich MW, Mackay CE, Jezzard P. Assessment of arterial arrival times derived from multiple inversion time pulsed arterial spin labeling MRI. Magn Reson Med. 2010 Mar;63(3):641-7. doi: 10.1002/mrm.22256. PMID 20146233
- [Result] MacIntosh BJ, Lindsay AC, Kylintireas I, Kuker W, Gunther M, Robson MD, Kennedy J, Choudhury RP, Jezzard P. Multiple inflow pulsed arterial spin-labeling reveals delays in the arterial arrival time in minor stroke and transient ischemic attack. AJNR Am J Neuroradiol. 2010 Nov;31(10):1892-4. doi: 10.3174/ajnr.A2008. Epub 2010 Jan 28. PMID 20110375
- [Result] MacIntosh BJ, McIlroy WE, Mraz R, Staines WR, Black SE, Graham SJ. Electrodermal recording and fMRI to inform sensorimotor recovery in stroke patients. Neurorehabil Neural Repair. 2008 Nov-Dec;22(6):728-36. doi: 10.1177/1545968308316386. Epub 2008 Sep 10. PMID 18784267
- See also: Sunnybrook Research website — http://www.sunnybrook.ca/research